CLINICAL TRIAL: NCT06628401
Title: A Comparison Between Different Approaches to Increase Fruit and Vegetable Intake and Influence Markers of Metabolic Health in Humans
Brief Title: Comparing Approaches to Increasing Fruit and Vegetable Intake and Their Influence on Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Courtney Neal (Other)
Collaborators: Newcastle University (Other); European Fruit Juice Association (AIJN) (Unknown)
Responsible Party: Sponsor-Investigator, Courtney Neal, Research Assistant, Newcastle University
Organization: Newcastle University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2792/48171; NU-019324 (Other Grant/Funding Number: The European Fruit Juice Association)
Record Dates: First submitted 2024-09-02; First posted 2024-10-08 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Health; Fruit and Vegetable Intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Control) (Placebo Comparator): Participants will be asked to maintain their habitual diet throughout the intervention. They will be provided with a brief document outlining the importance of a control group in research studies to maximise compliance. They will also receive £10/week vouchers during the intervention period and a further £60 on completion of the study to replicate voucher provision in the two intervention groups. Mimicking the voucher provision structure of the intervention groups will help to minimise participant drop out and will avoid any bias associated with differential financial remuneration between groups.
  Interventions: Behavioral: Educational information (Control)
- Group 2 (Whole F&V) (Active Comparator): Participants will be provided with educational material to increase their fruit and vegetable intake to meet 5-a-day guidelines via exclusive intake of whole fruits/vegetables . They will receive £10/week supermarket vouchers during the intervention period to support fruit/vegetable purchase. They will receive a further £60 on completion of the study.
  Interventions: Behavioral: Educational information (Increasing F&V intake)
- Group 3 (Whole F&V + Juice) (Experimental): Participants will be provided with educational material to increase fruit and vegetable intake to meet 5-a-day guidelines, with recommendations to consume one portion per day via fruit juice/smoothies. Participants will receive the same financial support as group 2.
  Interventions: Behavioral: Educational information (Increasing F&V intake + Juice)

INTERVENTIONS:
Behavioral: Educational information (Control) — Information packs will be developed for participants outlining the importance of a control group in research studies to maximise compliance. Participants will receive a £10 gift voucher weekly that they can spend at selected retailers of their choosing.
  Arms: Group 1 (Control)
Behavioral: Educational information (Increasing F&V intake) — Information packs will be developed to support participants in increasing their intake of whole fruits and vegetables, excluding fruit juice. The information packs will be developed using published guidance from the UK government, expert panels, and regulatory bodies. The packs will be co-developed with the public to ensure the guidance is appropriate for its target audience. Participants will also receive a £10 supermarket voucher weekly to purchase fruit and vegetables.
  Arms: Group 2 (Whole F&V)
Behavioral: Educational information (Increasing F&V intake + Juice) — Information packs will be developed to support participants in increasing their intake of whole fruits and vegetables, including fruit juice. The information packs will be developed using published guidance from the UK government, expert panels, and regulatory bodies. The packs will be co-developed with the public to ensure the guidance is appropriate for its target audience. Participants will also receive a £10 supermarket voucher weekly to purchase fruit and vegetables.
  Arms: Group 3 (Whole F&V + Juice)

SUMMARY:
This experimental study aims to evaluate the effects of different strategies for increasing fruit and vegetable intake and to see how these interventions influence markers of health in people aged 18-65 who currently consume fewer than 2 portions of fruit and vegetables a day.

The main questions it aims to answer are:

1. How does 5-a-day advice, with and without the inclusion of fruit juice, impact fruit and vegetable intake over a four-week period?
2. What are the acceptability and perceived ease of increasing fruit and vegetable intake with and without the inclusion of fruit juice in 5-a-day recommendations?
3. What are the effects of increasing fruit and vegetable intake with and without fruit juice on markers of metabolic health?

Researchers will answer these questions by comparing results from three groups of participants. All participants will provide a pre- and post-intervention blood sample, complete various questionnaires, and follow a four-week intervention that comprises educational material and a weekly £10 voucher. Over the course of the four weeks, they will report what they ate in a day on four different days.

The groups differ in the educational materials provided and where they can spend their voucher:

* Group 1 (Control) - information on the importance of including an experimental control in research and a weekly voucher to spend at a retailer of their choice,
* Group 2 (F&V) - information on 5-a-day advice (excluding fruit juice) and a weekly voucher to spend in a supermarket on F&V, and
* Group 3 (F&V + Juice) - information on 5-a-day advice (including fruit juice) and a weekly voucher to spend in a supermarket on F&V.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 65 years
* Currently consuming ≤2 portions of fruit and vegetables per day

Exclusion Criteria:

* Using high-dose vitamins, minerals or dietary supplements that could interfere with biomarker assessment of fruit and vegetable consumption
* Have a food sensitivity, allergy or other dietary restriction (e.g., following a weight loss diet) that would limit the ability to take part in the study
* Have a medical condition (e.g., diabetes or gastrointestinal disorders) that would limit the ability to take part in the study
* Currently pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Number of daily fruit and vegetable portions (from dietary recalls) | 4 weeks
  The number of daily portions of fruit and vegetables consumed (including fruit juice in group 3) will be determined by 4 x 24-hour dietary recalls using the validated dietary recall software Intake24 (Foster et al., 2019).

SECONDARY OUTCOMES:
Number of daily fruit and vegetable portions (from brief screening tool) | 4 weeks
  The 6-item fruit and vegetable screener module from the BRFSS (Behavioral Risk Factor Surveillance System; CDC, 2020) will be used as a secondary measure to capture self-reported fruit and vegetable intake pre- and post-intervention. Data will be compared against the more granular dietary data from Intake24, to evaluate agreement and suitability of this tools for use as an outcome measure in future fruit and vegetable-based interventions.
Concentration of plasma ascorbic acid | 4 weeks
  Prior to and following the intervention, participants will provide a fasted blood sample for determining objective biomarkers of fruit and vegetable intake. Concentration of plasma ascorbic acid (μmol/L), or vitamin C, will be measured via high-performance liquid chromatography (HPLC) using methods well-validated in our laboratory. These markers will help verify any participant-reported changes in fruit (including juice) and vegetable intake.
Concentration of serum carotenoids (lutein) | 4 weeks
  Prior to and following the intervention, participants will provide a fasted blood sample for determining objective biomarkers of fruit and vegetable intake. Concentration of the serum carotenoid lutein (μmol/L) will be measured via high-performance liquid chromatography (HPLC) using methods well-validated in our laboratory. These markers will help verify any participant-reported changes in fruit (including juice) and vegetable intake.
Concentration of serum carotenoids (zeaxanthin) | 4 weeks
  Prior to and following the intervention, participants will provide a fasted blood sample for determining objective biomarkers of fruit and vegetable intake. Concentration of the serum carotenoid zeaxanthin (μmol/L) will be measured via high-performance liquid chromatography (HPLC) using methods well-validated in our laboratory. These markers will help verify any participant-reported changes in fruit (including juice) and vegetable intake.
Concentration of serum carotenoids (beta-cryptoxanthin) | 4 weeks
  Prior to and following the intervention, participants will provide a fasted blood sample for determining objective biomarkers of fruit and vegetable intake. Concentration of the serum carotenoid beta-cryptoxanthin (μmol/L) will be measured via high-performance liquid chromatography (HPLC) using methods well-validated in our laboratory. These markers will help verify any participant-reported changes in fruit (including juice) and vegetable intake.
Concentration of serum carotenoids (lycopene) | 4 weeks
  Prior to and following the intervention, participants will provide a fasted blood sample for determining objective biomarkers of fruit and vegetable intake. Concentration of the serum carotenoid lycopene (μmol/L) will be measured via high-performance liquid chromatography (HPLC) using methods well-validated in our laboratory. These markers will help verify any participant-reported changes in fruit (including juice) and vegetable intake.
Concentration of serum carotenoids (alpha-carotene) | 4 weeks
  Prior to and following the intervention, participants will provide a fasted blood sample for determining objective biomarkers of fruit and vegetable intake. Concentration of the serum carotenoid alpha-carotene (μmol/L) will be measured via high-performance liquid chromatography (HPLC) using methods well-validated in our laboratory. These markers will help verify any participant-reported changes in fruit (including juice) and vegetable intake.
Concentration of serum carotenoids (beta-carotene) | 4 weeks
  Prior to and following the intervention, participants will provide a fasted blood sample for determining objective biomarkers of fruit and vegetable intake. Concentration of the serum carotenoid beta-carotene (μmol/L) will be measured via high-performance liquid chromatography (HPLC) using methods well-validated in our laboratory. These markers will help verify any participant-reported changes in fruit (including juice) and vegetable intake.
Concentration of metabolic health markers | 4 weeks
  Prior to and following the intervention, participants will provide a fasted blood sample to determine markers of metabolic health. The Nightingale metabolomic biomarker panel, assessed pre- and post-intervention using Nuclear Magnetic Resonance (NMR) spectroscopy, will be used to evaluate the impact of the intervention on markers of metabolic health.
Measure of depression symptom severity (PHQ-9) | 4 weeks
  The impact of the study interventions on symptoms of depression will be evaluated by administering the PHQ-9 questionnaire (a validated tool to measure levels of depression) pre- and post-intervention. Participants will provide information on the frequency with which they have been affected by depression-related symptoms (from not at all to nearly every day). There are four options for participants to select and each is associated with a score (not at all (0), several days (+1), more than half the days (+2), nearly every day (+3)). The sum of these scores indicates the level of depression severity (0-4 none/minimal; 5-9 mild anxiety; 10-14 moderate; 15 -19 moderately severe; 20-27 severe).
Measure of anxiety symptom severity (GAD-7) | 4 weeks
  The impact of the study interventions on anxiety symptoms will be evaluated by administering the GAD-7 questionnaire (a validated tool to measure levels of anxiety) pre- and post-intervention. Participants will provide information on the frequency with which they have been affected by anxiety-related symptoms. There are four options for participants to select, and each option is associated with a score (not at all (0), several days (+1), more than half the days (+2), and nearly every day (+3)). The sum of these scores indicates the level of anxiety (0-4 minimal; 5-9 mild anxiety; 10-14 moderate anxiety; greater than 15 severe anxiety).
Total number of gut symptoms (score) | 4 weeks
  Participants will complete the gut symptoms questionnaire (Winham and Hutchins, 2011) pre- and post-intervention. This involves responding to 4 close-ended questions (yes/no) enquiring about changes in the frequency of flatulence, stool frequency, stool consistency, or bloating frequency in the past week. The total number of symptoms the participant reported as having increased in the last week is their gut symptom score.
Change in flatulence symptoms | 4 weeks
  Participants will complete the gut symptoms questionnaire (Winham and Hutchins, 2011) pre- and post-intervention. One of these items is a close-ended question (yes/no) enquiring about changes in the frequency of flatulence in the past week. If participants report a change, they will be asked to indicate the direction (increase/decrease) and magnitude of change (from 1 = least change to 5 = greatest change on a 5-point likert scale).
Change in stool frequency | 4 weeks
  Participants will complete the gut symptoms questionnaire (Winham and Hutchins, 2011) pre- and post-intervention. One of these items is a close-ended question (yes/no) enquiring about changes in stool frequency in the past week. If participants report a change, they will be asked to indicate the direction (increase/decrease) and magnitude of change (from 1 = least change to 5 = greatest change on a 5-point likert scale).
Change in stool consistency | 4 weeks
  Participants will complete the gut symptoms questionnaire (Winham and Hutchins, 2011) pre- and post-intervention. One of these items is a close-ended question (yes/no) enquiring about changes in stool consistency in the past week. If participants report a change, they will be asked to indicate the direction (increase/decrease) and magnitude of change (from 1 = least change to 5 = greatest change on a 5-point likert scale).
Change in bloating frequency | 4 weeks
  Participants will complete the gut symptoms questionnaire (Winham and Hutchins, 2011) pre- and post-intervention. One of these items is a close-ended question (yes/no) enquiring about changes in bloating frequency in the past week. If participants report a change, they will be asked to indicate the direction (increase/decrease) and magnitude of change (from 1 = least change to 5 = greatest change on a 5-point likert scale).
Assessment of intervention acceptability | 4 weeks
  Acceptability of the interventions will be assessed post-study via a custom questionnaire, using 5-point visual analogue scales and informed by the Theoretical Framework of Acceptability (Sekhon et al., 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Oliver M Shannon, PhD, Principal Investigator — Newcastle University; Anthony Watson, PhD, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided